CLINICAL TRIAL: NCT01519349
Title: Phase I Clinical Intramuscular Gene Transfer of rAAV1.CMV.huFollistatin344 Trial to Patients With Becker Muscular Dystrophy and Sporadic Inclusion Body Myositis.
Brief Title: Follistatin Gene Transfer to Patients With Becker Muscular Dystrophy and Sporadic Inclusion Body Myositis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Collaborators: Parent Project Muscular Dystrophy (Other)
Responsible Party: Principal Investigator, Jerry R. Mendell, Director Center for Gene Therapy, Nationwide Children's Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NCH-696110
Record Dates: First submitted 2012-01-23; First posted 2012-01-26 (Estimated); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Becker Muscular Dystrophy; Sporadic Inclusion Body Myositis
Keywords: Becker muscular dystrophy; BMD; muscular dystrophy; inclusion body myositis; IBM; Follistatin
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Myositis, Inclusion Body; Muscular Dystrophies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort 1 (Experimental): Low Dose: 2E11 vg/kg of rAAV1.CMV.huFollistatin344 administered via intramuscular injection unilaterally to single quadriceps muscle (n=3, sIBM only)
  Interventions: Biological: rAAV1.CMV.huFollistatin344
- Cohort 2 (Experimental): Mid Dose: 3E11 vg/kg per quadriceps of rAAV1.CMV.huFollistatin344 administered via intramuscular injection bilaterally to both quadriceps muscles (n=6; 3 sIBM and 3 BMD)
  Interventions: Biological: rAAV1.CMV.huFollistatin344
- Cohort 3 (Experimental): Low Dose: 6E11 vg/kg per quadriceps of rAAV1.CMV.huFollistatin344 administered via intramuscular injection bilaterally to both quadriceps muscles (n=6; 3 sIBM and 3 BMD)
  Interventions: Biological: rAAV1.CMV.huFollistatin344

INTERVENTIONS:
Biological: rAAV1.CMV.huFollistatin344 — * First cohort - Low Dose: 2E11 vg/kg with single leg injection (n=3 sIBM)
  * Second cohort: 3E11 vg/kg per quad (n=3 sIBM; 3 BMD)
  * Third cohort: 6E11 vg/kg per quad (n=3 sIBM; 3 BMD)

SUMMARY:
The investigators are performing a gene therapy clinical trial in Becker muscular dystrophy (BMD) and sporadic inclusion body myositis (sIBM) patients. Both of these conditions have an important common feature: loss of ability to walk because of weakness of the thigh muscles. The investigators plan to do a gene therapy trial to deliver a gene to muscle called follistatin (FS344) that can build muscle size and strength. If successful, the investigators can increase the size of the thigh muscle and potentially prolong a patient's ability to walk. The gene will be carried into the muscle by a virus called adeno-associated virus (AAV). This virus occurs naturally in muscle and does not cause any human disease, setting the stage for its safe use in a clinical trial.

Presently there is no treatment that can reverse Becker muscular dystrophy or sporadic inclusion body myositis. Only supportive care is currently possible.

In this study, subjects with either of these diseases will have shots of the follistatin gene injected directly into thigh muscle on one (first cohort) or both legs (2nd and 3rd cohort). One hundred and eighty days following the gene delivery, the muscle will undergo biopsy to look closely at the muscle to see if the muscle fibers are bigger. Between the time of the gene transfer and the muscle biopsy, patients will be carefully monitored for any side effects of the treatment. This will include an MRI of the thigh muscle before treatment and at day 180 following treatment. Blood and urine tests, as well as physical examination will be done on the subjects during the screening visit and on days 0, 1, 2, 7, 14, 30, 60, 90, and 180 to make sure that there are no side effects from the gene injections. Sutures will be removed 2 weeks post-biopsy.

Additional blood samples will be collected at 9, 12, 18, and 24 months. Patients will be seen at the end of 1st and 2nd years for a physical exam, assessment of muscle strength and appropriate blood tests.

ELIGIBILITY:
Inclusion Criteria:

* All subjects [sIBM and BMD must be ambulatory and have identifiable atrophy of the quadriceps muscle with muscle weakness ≥2 standard deviations below predicted using quantitative muscle testing (maximum voluntary isometric strength testing), and difficulty getting out of chairs, climbing stairs, and getting up from the floor.
* sIBM patients include males and post-menopause females of any ethnic or racial group. Diagnosis of sIBM is based on previously published criteria that include distribution of weakness (knee extensor weakness, finger flexor weakness) and histological presence of inflammation and vacuolar myopathy. Patients with inflammation, vacuolar changes and intracellular amyloid deposits or 15/18nm filaments fulfill criteria irrespective of clinical features.
* BMD patients include adult males (>18yo) of any ethnic or racial group with proven mutation of dystrophin gene and continued ambulation after age 15 years old.
* Ability to cooperate for muscle testing
* Deficit in muscle strength greater than 2 standard deviation below age expectations
* Willingness of sexually active subjects with reproductive capacity (only male population) to practice reliable method of contraception until two negative sperm samples are obtained post gene transfer

Exclusion Criteria:

* Active viral infection
* History or evidence of active infection with hepatitis C, hepatitis A or B, or HIV
* Patients with any other cause of muscle weakness based on medical history and screening physical exam including: myopathy (other dystrophies, polymyositis, and dermatomyositis), neuropathy (from any cause), myasthenia gravis, and weakness related to degenerative joint disease of the spine.
* Ongoing immunosuppressive therapy or immunosuppressive therapy within 3 months of starting the trial (e.g. corticosteroids, cyclosporine, tacrolimus, methotrexate, cyclophosphamide, intravenous immunoglobulin, rituximab)
* Concomitant illness or requirement for chronic drug treatment that in the opinion of the PI creates unnecessary risks for gene transfer. Patients taking any of the following drugs will be excluded: drugs for treatment of myopathy or neuropathy or agents used to treat diabetes mellitus
* Knee or ankle contractures preventing proper muscle strength testing
* Patients with AAV1 neutralizing antibody titers ≥ 1:1600 as determined by ELISA immunoassay
* Patients with history of angina and patients with past history of myocardial infarction in the past 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-01; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Safety | 2 years
  Safety trial based on development of unacceptable toxicity defined as the occurrence of any Grade III or higher treatment-related toxicities.

SECONDARY OUTCOMES:
Muscle Function and Strength Testing | 2 years
  * Muscle function and strength:
  * MRI of quadriceps muscles (bilateral)
  * Muscle biopsies on quadriceps muscles (a muscle biopsy on one leg at baseline screening visit - except for cohort 1 - and the post gene transfer biopsy on the opposite leg at day 180)
  * Thigh circumference measurement at baseline and post-gene transfer follow up visits up to day 180 (prior to second biopsy)

CONTACTS AND LOCATIONS:
Overall Officials: Jerry R Mendell, M.D., Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

REFERENCES:
- [Background] Kota J, Handy CR, Haidet AM, Montgomery CL, Eagle A, Rodino-Klapac LR, Tucker D, Shilling CJ, Therlfall WR, Walker CM, Weisbrode SE, Janssen PM, Clark KR, Sahenk Z, Mendell JR, Kaspar BK. Follistatin gene delivery enhances muscle growth and strength in nonhuman primates. Sci Transl Med. 2009 Nov 11;1(6):6ra15. doi: 10.1126/scitranslmed.3000112. PMID 20368179
- [Background] Rodino-Klapac LR, Haidet AM, Kota J, Handy C, Kaspar BK, Mendell JR. Inhibition of myostatin with emphasis on follistatin as a therapy for muscle disease. Muscle Nerve. 2009 Mar;39(3):283-96. doi: 10.1002/mus.21244. PMID 19208403
- [Background] Miller TM, Kim SH, Yamanaka K, Hester M, Umapathi P, Arnson H, Rizo L, Mendell JR, Gage FH, Cleveland DW, Kaspar BK. Gene transfer demonstrates that muscle is not a primary target for non-cell-autonomous toxicity in familial amyotrophic lateral sclerosis. Proc Natl Acad Sci U S A. 2006 Dec 19;103(51):19546-51. doi: 10.1073/pnas.0609411103. Epub 2006 Dec 12. PMID 17164329
- [Result] Mendell JR, Sahenk Z, Malik V, Gomez AM, Flanigan KM, Lowes LP, Alfano LN, Berry K, Meadows E, Lewis S, Braun L, Shontz K, Rouhana M, Clark KR, Rosales XQ, Al-Zaidy S, Govoni A, Rodino-Klapac LR, Hogan MJ, Kaspar BK. A phase 1/2a follistatin gene therapy trial for becker muscular dystrophy. Mol Ther. 2015 Jan;23(1):192-201. doi: 10.1038/mt.2014.200. Epub 2014 Oct 17. PMID 25322757
- [Derived] Bian X, Snow ZK, Zinn CJ, Gowan CC, Conley SM, Bratulin AL, Elhusseiny KM, Miller J, Tchkonia T, Kirkland JL, Lerman LO, Hickson LJ. Activin A Antagonism with Follistatin Reduces Kidney Fibrosis, Injury, and Cellular Senescence-Associated Inflammation in Murine Diabetic Kidney Disease. Kidney360. 2025 Mar 28;6(8):1278-1291. doi: 10.34067/KID.0000000776. PMID 40152935
- See also: Click here for Center for Gene Therapy, The Research Institute at Nationwide Children's Hospital — http://www.nationwidechildrens.org/center-for-gene-therapy
- See also: Click here for Parent Project Muscular Dystrophy — http://www.parentprojectmd.org
- See also: Click here for The Myositis Association — http://www.myositis.org/